CLINICAL TRIAL: NCT02322879
Title: Protective Effects of Propylene Glycol in Daily Acetaminophen Dosing
Acronym: APAPII
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Harvard University (Other)
Responsible Party: Principal Investigator, Michael Ganetsky, Assistant Professor of Emergency Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2013P000070
Record Dates: First submitted 2014-10-22; First posted 2014-12-23 (Estimated); Results first posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Acetaminophen Toxicity
Keywords: Acetaminophen; Propylene glycol
MeSH Terms: interventions — WASH protein, Drosophila

STUDY DESIGN:
Intervention Model Description: Eligible subjects will then be randomized at a 1:1 ratio to receive either acetaminophen (APAP) or APAP + propylene glycol for 2 weeks (Treatment Period 1). At the end of the Treatment Period 1 subjects will enter the Wash-Out period for 2 weeks. Study subjects will then receive the alternative treatment for 2 weeks (Treatment Period 2). Overall, the maximum duration of treatment is approximately 6 weeks.
  RESPONDERS: Subjects whose transaminase levels rise to 3 times normal or greater during either of the Treatment Periods will be deemed responders and the intervention will cease.
  * If subjects are in the Treatment Period 1, they will enter the washout period and continue to return daily to ensure that liver function tests decline. After the 2 week washout-period, responders will cross over to Treatment Period 2.
  * If subjects are in the Treatment Period 2 phase, they will continue to return to the CRC and have their transaminases checked until they return to normal.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetaminophen first, then Acetaminophen + Propylene Glycol (Experimental): Subjects in this arm will receive 4 grams of solid acetaminophen formulation for two weeks, followed by a two week wash out period.
  Then, subjects will receive 4 grams of solid acetaminophen formulation in addition to 70 mg/kg/day of liquid propylene glycol for two weeks.
  The total study time is 6 weeks.
  Interventions: Drug: First Treatment Period; Other: Washout; Drug: Second Treatment Period
- Acetaminophen + Propylene Glycol first, then Acetaminophen (Experimental): Subjects in this arm will receive 4 grams of solid acetaminophen formulation in addition to 70 mg/kg/day of liquid propylene glycol for two weeks, followed by a two week wash out period.
  Then, subjects will receive 4 grams of solid acetaminophen formulation for two weeks.
  The total study time is 6 weeks.
  Interventions: Drug: First Treatment Period; Other: Washout; Drug: Second Treatment Period

INTERVENTIONS:
Drug: First Treatment Period — (duration: 14 days) Subjects will be randomized to receive either of the 2 interventions (4 grams of solid acetaminophen formulation for two weeks vs. 4 grams of solid acetaminophen formulation + 70 mg/kg/day of liquid propylene glycol)
Other: Washout — (duration: 14 days) At the end of the First intervention period all participants will enter a washout period.
Drug: Second Treatment Period — (duration: 14 days) At the end of the washout period, participants will receive the alternative intervention.

SUMMARY:
A purpose of this protocol is to is to compare the metabolites of the toxic bioactivating pathway after acetaminophen alone or acetaminophen followed by Propylene Glycol (PG) and to determine if it prevents the formation of the toxic metabolites of acetaminophen.

DETAILED DESCRIPTION:
The purpose of this protocol is to contribute to our overarching purpose, which is to determine if inhibiting the bioactivation of acetaminophen (APAP) can prevent liver injury, and to further describe the initiating mechanisms of APAP induced liver injury. APAP induced liver injury is caused by metabolism and/or the resulting metabolites when APAP undergoes reductive metabolism via the cytochrome P450 (CYP) system, principally via CYP 2E1. Inhibition of CYP 2E1 activity protects against toxicity in rodents and tissue culture. Our prior research indicates that inhibition of CYP 2E1 by administering a pediatric preparation of APAP containing Propylene Glycol (PG), a known CYP 2E1 inhibitor, results in reduced production of CYP 2E1 derived metabolites via competitive inhibition.

In this proposed protocol the investigators will provide therapeutic doses of APAP and a separately administered non toxic dose of PG over a two-week period to healthy subjects. 20-75% of healthy people who take therapeutic doses of APAP for 7-28 days will have an asymptomatic and subclinical rise in transaminase levels that will return to baseline without adverse effect or therapy. 3 The return to baseline occurs despite continued dosing of APAP.

A primary purpose is to determine if PG is, in fact, the substance in the liquid preparation responsible for the effect the investigators observed in the investigators initial study. A secondary purpose is to obtain plasma samples for secondary metabolomic analysis to elucidate the effect of CYP 2E1 inhibition.

Specific Aims

* 1 To demonstrate that co-administration of PG with APAP prevents the rise in AST/ALT expected in approximately one third of subjects following therapeutic dosing of APAP over days.
* 2 To show that PG administered with APAP reduces toxic P450-derived metabolite production following therapeutic APAP administration.
* 3 To obtain plasma samples to undergo metabolomic and other analyses to determine the effects of CYP 2E1 inhibition in the setting of APAP administration.
* 4 To undergo metabolomic analyses on the day LFT's peak to determine differences in metabolomics parameters between subjects receiving propylene glycol plus acetaminophen versus just acetaminophen alone.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers ages 20-40
* Patients not taking any chronic medications

Exclusion Criteria:

* Any history of liver disease
* Frequent alcohol use (2 or more drinks more than 4 times per week)
* Pregnant women
* Chronic medical condition requiring daily pharmacotherapy or the use of any daily prescription medications.
* Unable to provide informed consent

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2013-05; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Salhanick, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
We plan to publish the data in near future but there is no plan on sharing the individual participant data

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After responding to the internet or print advertisement, prospective subjects were scheduled for a screening visit at the Harvard Catalyst Clinical Research Center (CRC) at BIDMC between May 2013 and August 2016. In all participants, consent was obtained prior to initiating any screening evaluation.
Groups:
- Acetaminophen First, Then Acetaminophen + Propylene Glycol: Participants in this arm received 4 grams of solid acetaminophen formulation for two weeks, followed by a two week wash out period.
  Then, subjects received 4 grams of solid acetaminophen formulation in addition to 70 mg/kg/day of liquid propylene glycol for two weeks.
- Acetaminophen + Propylene Glycol First, Then Acetaminophen: Participants in this arm received 4 grams of solid acetaminophen formulation in addition to 70 mg/kg/day of liquid propylene glycol for two weeks, followed by a two week wash out period.
  Then, subjects received 4 grams of solid acetaminophen formulation for two weeks.
Period: First Intervention
Arm/Group | Acetaminophen First, Then Acetaminophen + Propylene Glycol | Acetaminophen + Propylene Glycol First, Then Acetaminophen
Started | 11 | 10
Completed | 10 | 10
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0
Period: Washout
Arm/Group | Acetaminophen First, Then Acetaminophen + Propylene Glycol | Acetaminophen + Propylene Glycol First, Then Acetaminophen
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Acetaminophen First, Then Acetaminophen + Propylene Glycol | Acetaminophen + Propylene Glycol First, Then Acetaminophen
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetaminophen First, Then Acetaminophen + Propylene Glycol | Acetaminophen + Propylene Glycol First, Then Acetaminophen | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Full Range); unit: years] | 28.6 [21 to 37] | 29.8 [24 to 37] | 29.2 [21 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Rise in Plasma Transaminases: Proportion of Responders.
Description: Blood tests to monitor Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) were obtained on every visit prior dosing. ALT and AST were analyzed on a Roche Cobas c501 chemistry module at BIDMC. Responders was defined as peak ALT increased 2x baseline (average of first 3 days)
Time Frame: Daily during the treatment periods (D1-D14 and D29 to 42)
Measure: Count of Participants; unit: Participants
Groups:
- Acetaminophen: Participants received 4 grams of solid acetaminophen formulation for two weeks
- Acetaminophen + Propylene Glycol: Participants received 4 grams of solid acetaminophen formulation in addition to 70 mg/kg/day of liquid propylene glycol for two weeks
Arm/Group | Acetaminophen | Acetaminophen + Propylene Glycol
Number analyzed (Participants) | 21 | 20
Participants | 6 | 8
Statistical Analysis 1: Comparison: Acetaminophen vs Acetaminophen + Propylene Glycol; Test type: Superiority; p = 0.59, Chi-squared

ADVERSE EVENTS:
Time Frame: During Participation in the study (6 weeks)
Description: Adverse events were be monitored at every by trained investigators at the Harvard-Thorndike Clinical Research Center at Beth Israel Deaconess Medical Center. Additionally, study participants were instructed to contact the study team for any symptoms out of the ordinary.
Arm/Group | Acetaminophen | Acetaminophen + Propylene Glycol
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/21 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No